CLINICAL TRIAL: NCT00150059
Title: Efficacy and Safety of Pimecrolimus Cream 1% in Patients ≥ 3 Months of Age With Mild or Moderate Atopic Dermatitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASM981CPH01
Record Dates: First submitted 2005-09-07; First posted 2005-09-08 (Estimated); Last update posted 2008-02-15 (Estimated); Status verified 2008-02

CONDITIONS: Atopic Dermatitis
Keywords: atopic dermatitis, eczema, mild to moderate, children, IGA
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — pimecrolimus

INTERVENTIONS:
Drug: Pimecrolimus Cream 1%
  Other Names: Elidel

SUMMARY:
To evaluate the efficacy and safety of pimecrolimus cream 1% in its registered indication (treatment of patients > 3 months of age with mild to moderate atopic dermatitis)

This study is not enrolling patients in the United States.

ELIGIBILITY:
The patient population must consist of male or female outpatients, age ≥3 months old with mild to moderate atopic dermatitis (IGA ≥ 1). Exclusion criteria are pregnancy, having active viral infections at the site(s) of treatment, presenting with systemic malignancy or active lymphoproliferative diseases/disorders, receiving phototherapy or immunosuppressive therapy, having used tacrolimus ointment and known allergy or hypersensitivity.

Min Age: 3 Months | Sex: All
Age Groups: Child, Adult, Older Adult
Dates: Start 2004-12; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Investigator Global Assessment (IGA) score for the whole body and for the face only.
Pruritus (itch) severity assessments, and patient's self-assessment of disease control at the start of study and on day 7, 30 and 90 after treatment initiation.
Safety assessed by adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Healthcare Philippines, Study Chair — Novartis Pharmaceuticals
Locations (1):
- This study is not being conducted in the United States, Investigative Site, Philippines